CLINICAL TRIAL: NCT06683638
Title: Daily Doxycycline for Early Syphillis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Travis J Hunt, Clinician Researcher, Division of Allergy and Infectious Diseases, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021340
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Syphilis
Keywords: syphilis; doxycycline
MeSH Terms: conditions — Syphilis | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: This study will enroll one prospective arm of 15 persons. To contextualize the finding, the investigators will separately determine point-estimates of 6-month treatment response to standard of care regimens in the sexual health program using de-identified retrospective cohorts of 60 persons each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doxycycline 200mg daily for 14 days (Experimental): Participants diagnosed with early syphilis (primary, secondary, or early latent) with an RPR of 1:4 or greater will receive doxycycline 200mg daily to treat syphilis. Exclusions include pregnant persons, persons under 18 years of age, and persons on doxy PEP. During the two weeks of treatment, participants will perform oral and rectal swabs for syphilis, returned at the end of the 2 weeks by mail. Participants will submit brief online surveys twice over the two weeks of treatment. Repeat blood tests for syphilis, reactive plasma reagin (RPR), will be done at follow-up visits at 3 and 6 months to monitor serological response. Participants with response at the 3-month visit will not need to come to a 6-month visit.
  Interventions: Drug: Doxycycline 200mg daily for 14 days

INTERVENTIONS:
Drug: Doxycycline 200mg daily for 14 days — Doxycycline will be taken as a single dose of 200mg daily, rather than the current CDC-recommended 100mg twice daily regimen for early syphilis. The duration will still be 14 days of therapy.

SUMMARY:
The goal of this clinical trial is to learn if doxycycline taken as 200mg daily for 14 days is effective to treat early stage syphilis. This is different from how doxycycline is typically used for syphilis because the full doxycycline dose will be taken at the same time of day, rather than split up into a twice daily regimen. Lab data support that taking the medication as a single daily dose should be effective as treatment, but it has not been studied clinically. The main question this study aims to answer is:

Is doxycycline taken as a single daily dose of 200mg for 14 days an effective treatment for early syphilis based on a combined outcome of clinical improvement and blood test improvement?

Participants will:

1. Take doxycycline 200mg daily for 14 days
2. Submit oral and rectal swabs that test for syphilis bacteria every other day for 2 weeks, returned by mail
3. Complete 2 brief online surveys over the first 2 weeks
4. Return to the clinic for an interview and blood draw every 3 months for a maximum of 3 study visits, including the first visit

The investigators will compare the percentage of participants in the study who have response to treatment by 6 months to that of persons who have received standard (CDC-recommended) regimens. To do this, the investigators will calculate response percentage estimates following a shot of long-acting penicillin or 14 days of doxycycline 100mg twice daily from 60-person samples from the sexual health program's records.

DETAILED DESCRIPTION:
This is an open-label prospective cohort of 15 participants diagnosed with early syphilis treated with doxycycline 200mg daily for 14 days. The outcome of interest is clinical improvement and fourfold decline in RPR by 6 months. This study will include rectal and oropharyngeal sampling with syphilis transcription-mediated amplification (TMA), every other day for the 14-day course, returned by mail. The investigators will obtain 6-month point estimates for cure following single-dose intramuscular benzathine penicillin G or 14 days of doxycycline 100mg twice daily in retrospective cohorts of 60 persons. The investigators will use binomial exact calculation with an alpha of 0.05, two-tailed, to create a point estimates of percent cure. The investigators will report TMA positivity descriptively.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of syphilis (primary or secondary) or laboratory-confirmed early latent syphilis. Specifically: This will include persons meeting any one of the following criteria:

1. Clinical diagnosis of primary syphilis (based on the presence of a chancre) and either a positive qualitative RPR in the absence of a prior positive RPR on their most recent serological test for syphilis or a positive darkfield microscope exam of material taken from a chancre, OR
2. Clinical diagnosis of secondary syphilis with a positive qualitative RPR in the absence of a prior positive RPR on their most recent serological test for syphilis, OR
3. A laboratory-confirmed diagnosis of early latent syphilis within one month (i.e. <31 days prior).

Exclusion Criteria:

1. age under 18
2. persons with evidence of neurosyphilis (including ocular and otic syphilis) or tertiary syphilis
3. persons who are unable to give informed consent
4. persons deemed by the study investigators to be unable to complete study follow-up visits
5. persons with an allergy to doxycycline
6. pregnant persons
7. persons with HIV who report that they are off antiretroviral medication or that they are not virologically suppressed
8. persons with other known forms of immunosuppression (e.g., persons taking systemic immunosuppressant drugs, persons with primary immunodeficiencies)
9. persons taking medications that would interact with doxycycline
10. persons whose initial RPR is lower than 1:4
11. persons currently prescribed doxy PEP
12. breastfeeding persons

Persons whose initial laboratory serological tests do not confirm the diagnosis of syphilis with an RPR of 1:4 or higher will be informed that they do not meet study criteria and advised to discontinue doxycycline 200mg once daily. Their subsequent treatment will be based on the judgement of non-research, clinical staff in the clinic and reflect shared decision making between clinical providers and their patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Composite clinical and serological response | 6 months
  Clinical response and serological response will be aggregated to arrive at one reported value, a binary outcome of "yes" (1) or "no" (0).
  Clinical response equates to resolution of clinical symptoms of syphilis the participants presented with, such as rash or chancre, without the development of new symptoms of syphilis. Resolution will be marked as "yes" or "no".
  Serological response equates to a fourfold decrease in RPR compared to the presenting RPR titer by 6 months. Resolution will be marked as "yes" or "no".
  Thus, to generate the composite response outcome, participants with outcomes of "yes" for both clinical response and serological response will qualify as a binary outcome of "yes" (1) . Participants who do not have outcomes of "yes" for both clinical response and serological response will qualify as a binary outcome of "no" (0).

CONTACTS AND LOCATIONS:
Overall Officials: Travis Hunt, MD, Principal Investigator — University of Washington
Locations (1):
- Public Health Sexual Health Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT06683638/ICF_001.pdf